CLINICAL TRIAL: NCT01673984
Title: A Phase IV, Randomised, Open-label, Multi-centre Study to Assess the Impact on Disease Control, Safety, Patient and Clinician Experience of Changing Patients With Advanced Prostate Cancer From a 3-monthly LHRH Agonist to 6-monthly Injections of Decapeptyl® SR 22.5 MG
Brief Title: GP Extended Action Triptorelin
Acronym: GREAT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was discontinued prematurely by the sponsor due to non-medical reasons
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-97-52014-181; 2011-004213-16 (EudraCT Number)
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Results first posted 2015-09-29 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decapeptyl® SR 22.5mg (Triptorelin) (Experimental)
  Interventions: Drug: Decapeptyl® SR 22.5mg
- Current 3-monthly LHRH agonist (Active Comparator): One of the following: Decapeptyl® SR 11.25mg (Triptorelin), Prostap® 3 DCS 11.25mg, Zoladex® LA 10.8mg
  Interventions: Drug: Decapeptyl® SR 11.25mg; Prostap® 3 DCS 11.25mg; Zoladex® LA 10.8mg

INTERVENTIONS:
Drug: Decapeptyl® SR 22.5mg — 22.5mg, intramuscular injection, given on day 1 / month 0 & month 6 (+/- 7 days).
  Other Names: Triptorelin
  Arms: Decapeptyl® SR 22.5mg (Triptorelin)
Drug: Decapeptyl® SR 11.25mg; Prostap® 3 DCS 11.25mg; Zoladex® LA 10.8mg — For Decapeptyl® SR 11.25mg: 11.25 mg, intramuscular injection For Prostap® 3 DCS 11.25mg: 11.25mg, depot injected subcutaneously For Zoladex® LA 10.8mg: 10.8mg, depot injected subcutaneously into anterior abdominal wall
  Other Names: Triptorelin
  Arms: Current 3-monthly LHRH agonist

SUMMARY:
The purpose of this study is to demonstrate that treatment with a 6-monthly injection of hormone therapy is as good and as well tolerated as the standard 3-monthly hormone therapy injections available for treating prostate cancer. The study will also aim to answer whether both doctors and patients would prefer treatment with a 6-monthly injection rather than injections every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written (personally signed and dated) informed consent before completing any study related procedure.
* Patients must be 18 years old or over.
* Patients must have a documented diagnosis of locally advanced or metastatic prostate cancer suitable for hormonal treatment
* Patients must be medically castrated with serum testosterone ≤ 0.5ng/mL
* Patients must have received at least two injections of a 3- monthly LHRH agonist by the time of the screening tests
* Patients must be stable on a 3-monthly LHRH agonist injection with stable PSA levels between screening and baseline (i.e. the baseline value must either be lower or less than 25% higher than the Screening value or if ≥25% higher, ≤0.5ng/mL higher than the screening value).

In addition:

* For patients with locally advanced prostate cancer (M0), LHRH agonist injection (any formulation) must have been initiated within the last 3 years from Baseline,
* For patients with metastatic prostate cancer (M+) and a Gleason score

  ≤ 7, LHRH agonist injection (any formulation) must have been initiated within the last 2 years from Baseline,
* For patients with metastatic prostate cancer (M+) and a Gleason score > 7, LHRH agonist injection (any formulation) must have been initiated within the last 12 months from Baseline.
* Patients must have an estimated life expectancy of at least twelve months according to the investigator's assessment.

Exclusion Criteria:

* Patients have had previous surgical castration or present any concomitant condition which could compromise the objectives of the study and/or preclude the protocol-defined procedures (e.g. severe medical conditions, brain metastases, psychiatric disorders, active or uncontrolled infection, known pituitary disease).
* Patients are, in the opinion of the investigator, unable to comply fully with the protocol and the study instructions.
* Patients have received investigational drug(s) or treatment(s) within 30 days prior to study entry or will require a concurrent treatment with any other experimental drugs or treatments or present any concomitant condition which could compromise the objectives of the study and/or preclude the protocol-defined procedures (e.g. severe medical conditions, brain metastases, psychiatric disorders, active or uncontrolled infection, known pituitary disease).
* Patients have had a diagnosis of any other cancer without a history of stability/remission within five years of screening, with the exception of non-metastatic basal cell carcinoma.
* Patients currently taking additional anti-androgen therapy as part of an active hormonal control therapy.
* Patients scheduled to receive palliative radiotherapy during the course of the study.
* Patients receiving an LHRH agonist as neo-adjuvant to radiotherapy or adjuvant to radiotherapy.
* Patients receiving LHRH agonist as adjuvant to surgery.
* Patients scheduled to undergo radical prostatectomy during the course of the study.
* Patients with known hypersensitivity to LHRH agonists, their analogues or any or any other component of the products to be administered.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (35):
- United Kingdom (35):
  - The Crouch Oak Family Practice, Addlestone
  - Dr Carter & Partners, Ashford
  - Westongrove Research Centre, Aston Clinton Surgery, Aylesbury
  - Clinical Research Unit, Oldfield Surgery, Bath
  - Clinical Research Unit, The Pulteney Practice, Bath
  - St James' Surgery, Bath
  - Waterloo Medical Centre, Blackpool
  - Woolpit Health Centre, Bury St Edmunds
  - Cossington House Surgery, Canterbury
  - Research Office, Avondale Surgery, Chesterfield
  - Clinical Research Dept., Rowden Surgery, Chippenham
  - Clinical Research Unit, Hathaway Medical Centre, Chippenham
  - The Porch Surgery, Corsham
  - Pound Hill Surgery, Crawley
  - The Medical Centre, East Horsley
  - Burbage Surgery, Hinckley
  - The Portmill Surgery, Hitchin
  - Townhead Surgery, Irvine
  - Mortimer Surgery, Mortimer Common
  - Kiltearn Medical Centre, Nantwich
  - Danes Camp Surgery, Northampton
  - Kingsthorpe Medical Centre, Northampton
  - Cape Cornwall Surgery, Penzance
  - The Alverton Practice, Penzance
  - Wansford & Kings Cliffe Practice, Wansford Surgery, Peterborough
  - Knowle House Surgery, Plymouth
  - The Rame Group Practice, Plymouth
  - Sherbourne Medical Centre, Royal Leamington Spa
  - Ashfields Primary Care Centre, Sandbach
  - Brannel Surgery, St Austell
  - Sunbury Health Centre Group Practice, Sunbury-on-Thames
  - Adcroft Surgery, Trowbridge
  - Sheepcot Medical Centre, Watford
  - Albany House Medical Centre, Wellingborough
  - Woosehill Medical Centre, Wokingham

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 subjects screened and 27 subjects were enrolled. Following enrollment, 21 patients were randomised before the study was prematurely discontinued.
Groups:
- Current 3-monthly LHRH Agonist: One of the following: Decapeptyl® SR 11.25mg, Prostap® 3 DCS 11.25mg, Zoladex® LA 10.8mg
  Decapeptyl® SR 11.25mg; Prostap® 3 DCS 11.25mg; Zoladex® LA 10.8mg: For Decapeptyl® SR 11.25mg: 11.25 mg, intramuscular injection For Prostap® 3 DCS 11.25mg: 11.25mg, depot injected subcutaneously For Zoladex® LA 10.8mg: 10.8mg, depot injected subcutaneously into anterior abdominal wall
Period: Overall Study
Arm/Group | Decapeptyl® SR 22.5mg | Current 3-monthly LHRH Agonist
Started | 14 | 7
Completed | 4 | 1
Not Completed | 10 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Study termination | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decapeptyl® SR 22.5mg | Current 3-monthly LHRH Agonist | Total
Number analyzed (Participants) | 14 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.2 (5.4) | 78.7 (9.3) | 77.7 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 7 | 21
Employment status/Occupation [Number; unit: participants]
  Employed | 2 | 1 | 3
  Retired | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Biochemical Castration
Description: Patients with serum total testosterone (STT) level lower than 0.5 ng/mL after 6 months of treatment.
Time Frame: 6 months
Population: Analysis based on intent-to-treat (ITT) population comprised of 21 patients.
Measure: Number; unit: percentage of participants
Arm/Group | Decapeptyl® SR 22.5mg | Current 3-monthly LHRH Agonist
Number analyzed (Participants) | 14 | 7
percentage of participants | 92.9 | 100

2. Secondary Outcome: Percentage of Participants Maintaining Biochemical Castration After 12 Months of Treatment.
Description: Patients with serum total testosterone (STT) level lower than 0.5 ng/mL, 12 months after randomisation..
Time Frame: 12 months
Population: Analysis based on the number of subjects with a valid value in the ITT population comprised of 21 patients.
Measure: Number; unit: percentage of participants
Arm/Group | Decapeptyl® SR 22.5mg | Current 3-monthly LHRH Agonist
Number analyzed (Participants) | 9 | 4
percentage of participants | 22.2 | 25.0

3. Secondary Outcome: Percentage of Participants Demonstrating Stable Prostate-specific Antigen (PSA) Levels
Description: Stable PSA level was noted as value either lower or less than 25% higher than the baseline value, or PSA value ≤0.5 ng/mL higher than the baseline value, if value ≥25% higher than the baseline value.
Time Frame: 6 and 12 months
Population: Analysis based on number (n) of patients with a valid value in the intent-to-treat (ITT) population which comprised of 21 patients.
Measure: Number; unit: percentage of participants
Arm/Group | Decapeptyl® SR 22.5mg | Current 3-monthly LHRH Agonist
Number analyzed (Participants) | 13 | 7
percentage of participants
  6 months (n = 13, 7) | 84.6 | 100
  12 months (n = 2, 1): number analyzed (Participants) | 2 | 1
  12 months (n = 2, 1) | 50 | 100

4. Secondary Outcome: Change From Baseline in Quality of Life Using EuroQol 5 Dimensions 5 Levels [EQ-5D-5L] Questionnaire.
Description: The EQ-5D-5L questionnaire consisted of a description of raw data which comprised of five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension had five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The visual analogical scale of the EQ-5D-5L questionnaire was numbered from 0 to 100 (0 meaning the worst health the patient can imagine and 100 the best health the patient can imagine).
Time Frame: Baseline and Month 12
Population: Analysis based on the number of subjects with a valid value in the ITT population which comprised of 21 patients.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Decapeptyl® SR 22.5mg | Current 3-monthly LHRH Agonist
Number analyzed (Participants) | 3 | 2
units on a scale | 71.7 [40.4 to 102.9] | 70.0 [-57.1 to 197.1]

5. Secondary Outcome: Change From Baseline in Patient Satisfaction With Medication Using Treatment Satisfaction Questionnaire for Medication (TSQM Version II)
Description: TSQM comprised of four dimensions: effectiveness, side effects, convenience and overall global satisfaction. Each score ranged from 0 to 100. For effectiveness, convenience and overall global satisfaction scores, 0 indicated an extreme dissatisfaction and 100 indicated an extreme satisfaction. For side effects score, 0 indicated an extreme dissatisfaction and 100 indicated no dissatisfaction at all.
Time Frame: 6 and 12 month
Population: Analysis based on the number (n) of subjects with a valid value in each arm of the ITT population which comprised of 21 patients.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Decapeptyl® SR 22.5mg | Current 3-monthly LHRH Agonist
Number analyzed (Participants) | 14 | 7
units on a scale
  Baseline to 6 months - Effectiveness (n= 13, 7): number analyzed (Participants) | 13 | 7
  Baseline to 6 months - Effectiveness (n= 13, 7) | 3.2 [-12.5 to 18.9] | 13.1 [-10.8 to 37.0]
  Baseline to 12 months - Effectiveness (n= 3, 2): number analyzed (Participants) | 3 | 2
  Baseline to 12 months - Effectiveness (n= 3, 2) | -33.3 [-74.7 to 8.1] | -12.5 [-383.1 to 358.1]
  Baseline to 6 months - Side Effects (n= 13, 7): number analyzed (Participants) | 13 | 7
  Baseline to 6 months - Side Effects (n= 13, 7) | -2.6 [-12.9 to 7.8] | 4.8 [-6.0 to 15.5]
  Baseline to 12 months - Side Effects (n= 3, 2): number analyzed (Participants) | 3 | 2
  Baseline to 12 months - Side Effects (n= 3, 2) | -25.0 [-115.2 to 65.2] | 12.5 [-146.3 to 171.3]
  Baseline to 6 months - Convenience (n= 13, 7): number analyzed (Participants) | 13 | 7
  Baseline to 6 months - Convenience (n= 13, 7) | 4.7 [-6.3 to 15.7] | 2.0 [-9.8 to 13.7]
  Baseline to 12 months - Convenience (n= 3, 2): number analyzed (Participants) | 3 | 2
  Baseline to 12 months - Convenience (n= 3, 2) | -1.9 [-36.6 to 32.9] | 2.8 [-103.1 to 108.7]
  Baseline to 6months -Global Satisfaction(n= 12, 6): number analyzed (Participants) | 12 | 6
  Baseline to 6months -Global Satisfaction(n= 12, 6) | -0.7 [-15.9 to 14.5] | -4.2 [-11.5 to 3.2]
  Baseline to 12months -Global Satisfaction(n= 2, 2): number analyzed (Participants) | 2 | 2
  Baseline to 12months -Global Satisfaction(n= 2, 2) | -12.5 [-171.3 to 146.3] | 4.2 [-48.8 to 57.1]

6. Secondary Outcome: Patient Satisfaction With Treatment.
Description: Using a non-validated study-specific descriptive Likert-type scale (with no units) comprising a simple six-question patient questionnaire.
Time Frame: Month 12
Population: No participant analysis as no data was collected due to low number of participants recruited in the study.
Arm/Group | Decapeptyl® SR 22.5mg | Current 3-monthly LHRH Agonist
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants Who Changed Injection Frequency After Completion of the Study
Time Frame: Month 12
Population: Analysis based on the number of subjects with a valid value in the ITT population which comprised of 21 patients.
Measure: Number; unit: percentage of participants
Arm/Group | Decapeptyl® SR 22.5mg | Current 3-monthly LHRH Agonist
Number analyzed (Participants) | 5 | 3
percentage of participants | 80 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Decapeptyl® SR 22.5mg | Current 3-monthly LHRH Agonist
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/7
Other Adverse Events (participants affected / at risk) | 12/14 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decapeptyl® SR 22.5mg (N=14) | Current 3-monthly LHRH Agonist (N=7)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decapeptyl® SR 22.5mg (N=14) | Current 3-monthly LHRH Agonist (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Suprapubic pain (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Serum ferritin increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No